CLINICAL TRIAL: NCT01116999
Title: Clinical Comparison of Direct Pharyngoscopic Tracheal Intubation Technique With Light-guided Tracheal Intubation
Brief Title: Retrograde Light Target Tracheal Intubation Technique:Clinical Comparison With Direct Pharyngoscopic Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, Yang Tao, Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital, Second Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19781007
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Tracheal Intubation Morbidity
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tracheal intubation (Experimental)
  Interventions: Procedure: light guided tracheal intubation

INTERVENTIONS:
Procedure: light guided tracheal intubation — Tracheal intubation light guided technique.
  Other Names: intubation

SUMMARY:
The investigators hypothesise that, for novices, light guided tracheal intubation will improve the time and success rate of this clinical skill compared to standard direct tracheal intubation.

DETAILED DESCRIPTION:
The experiment was conducted under the close supervision of the coaching anesthesiologists in several stages.

The training stage: First of all, the operators received training with respect to the theories and principles of airway management, including techniques of bag-mask ventilation, Direct laryngoscopy and tracheal intubation and light-guided and tracheal intubation until they had a good master about the theoretical background, technical risks and indications of the two techniques. Then, they had to receive manikin training of the two techniques on the Airway Management Trainer. Exposure of the glottis(EG)/tracheal intubation(TI) training would be continued before they were able to use both techniques to complete three consecutive cases of Exposure of the glottis/tracheal intubation operation successfully on the manikin trainer within 120 seconds (s) at a time.

20 medical workers were assigned to perform TI within 120s with either Direct laryngoscopy TI or light-guided TI technique, which was selected randomly and then converted to the alternative one until they complete 5 cases with each of the two techniques. The time of EG started from mouth opening of the patient to the exposure of the glottis. The time of TI also started from mouth opening of the patient to the completion of inserting the tracheal guide to the tracheal and sealing it with cuff inflation. The EG time, Cormack-Lehane (C&L) grades, TI time, one-time success rate, and the overall success rate in using the two TI techniques were recorded.

The patient was laid in a supine position, with the head laid on a 7cm-high pillow for the sake of stability. The peripheral vein was accessed routinely and connected to a standard monitor for electrocardiography (ECG), SpO2 and noninvasive blood pressure (BP). Sufficient oxygen inhalation was initiated for > 3min before induction of general anesthesia with midazolam, propofol, fentanyl and rocuronium bromide. The anesthesiologist was not allowed to give any instruction and suggestion or assistance to the operator during the whole process. The coaching anesthesiologist supervised the whole TI process closely. Should any hidden risk occur or the TI exceed the required time of the experiment, the TI attempt of the operator would be terminated and replaced by the anesthesiologist in order to ensure patients' safety: TI exceeded 120s; Attempt of TI exceeded 2 times; SpO2 decreasing to below 95%; appearance of unstable hemodynamic situations (mean BP or HR fluctuating by more than 25% of the baseline value); or occurrence of airway injury as evidenced by stained blood on the Macintosh Blade. Any patient with C&L grade III~IV as discovered by the anesthesiologist during TI would be excluded from the present study and replaced by anther patient to re-start the experiment. A 7.0- or 7.5-mm-ID endotracheal tube was used as the guide according to the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* age range 18~55 years
* general anesthesia
* ASA I~II
* Mallampati Score grade I~II
* thyromental distance ≥6cm
* mouth-open ≥3cm
* body mass index (BMI) ≤30kg/m2

Exclusion Criteria:

* neck and maxillofacial surgeries
* temporomandibular joint (TMJ) disease
* potential risks for regurgitation and pulmonary aspiration
* in pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Ease to intubate (time and success rate required to perform intubation) | Within 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, MD, Study Director — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University; Jiong Hou, MD, Study Director — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University; Xiaoming Deng, Professor, Study Director — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University; Xu Zhang, MD, Principal Investigator — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University; Wen Ni, MD, Principal Investigator — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University; Xiaoyan Zhu, MD, Principal Investigator — Second Military Medical University; Jinbao Li, MD, Principal Investigator — Department of Anesthesiology and Cirtical Care Medicine, Changhai Hospital Affiliated to Second Military Medical University
Locations (1):
- Changhai Hospital Affiliated to Second Military Medical University, Shanghai, Shanghai Municipality, China